CLINICAL TRIAL: NCT07028216
Title: Mindful Self-Compassion for Anxiety and Depression: A Randomized Comparison of In-Person Versus Videoconference Delivery
Brief Title: Mindful Self-compassion for Anxiety and Depression: Impact of Delivery Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Elizabeth Hoge, Professor of Psychiatry, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00005863-1
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia; Major Depressive Disorder; Persistent Depressive Disorder (Dysthymia)
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Depressive Disorder, Major; Dysthymic Disorder

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study investigator will be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person MSC (Experimental): Mindful Self-Compassion (MSC) is a weekly class given for 8 weeks. The individual classes last about 2 hours each. The class is provided in a group setting.
  Interventions: Behavioral: Mindful Self-Compassion
- Video-conference MSC (Active Comparator): Mindful Self-Compassion (MSC) is a weekly class given for 8 weeks. The individual classes last about 2 hours each. The class is provided in a video-conference group setting.
  Interventions: Behavioral: Mindful Self-Compassion

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — The course teaching mindfulness meditation skills relevant to cultivating self-compassion.

SUMMARY:
The study will compare the delivery of an 8-week Mindful Self-Compassion training, in-person against video-conference, on anxiety and depression symptom severity in patients with diagnosed anxiety disorders (generalized anxiety disorder, social anxiety disorder, and panic disorder) or major depressive disorder or dysthymia.

DETAILED DESCRIPTION:
Anxiety disorders, such as generalized anxiety disorder, social anxiety disorder, and panic disorder, and depressive disorders result in significant distress, impairment in social and occupational functioning and increased risk for suicide. While there are medication and psychotherapy treatment options, they can sometimes be difficult to access and may be ineffective for a proportion of the population. Also, many patients are reluctant to take psychiatric medication, and many prefer to avoid psychiatric care altogether due to stigma or distrust of medical care settings such as a psychiatry clinic. Mindfulness meditation training can be provided outside of a medical care setting and may be more acceptable and feasible for some patients.

One way that mindfulness meditation may provide unique benefits for anxiety and depression is through decreasing self-judgment and increasing self-compassion. Research has shown that people with anxiety disorders, for example, have lower levels of self-compassion than people without anxiety. This is consistent with theories about the development and phenomenology of anxiety disorders, which are characterized as having high levels of self-criticism. Mindfulness-based interventions have been shown to improve self-compassion and self-acceptance.

In this study, patients with anxiety disorders or depression will be randomized to either an in-person 8-week class called Mindful Self-Compassion training or a video-conference 8-week class called Mindful Self-Compassion.

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary anxiety disorder (social anxiety disorder, generalized anxiety disorder, panic disorder, or agoraphobia) or major depressive disorder, current
* Must score low on self-compassion, as measured by the self-compassion scale
* Must understand study procedure and willing to participate in all testing visits, and treatment as assigned
* Must be able to give informed consent to the study procedures

Exclusion Criteria:

* Comorbid psychiatric disorder other than anxiety or depression, such as psychotic disorder, obsessive compulsive disorder, eating disorders (i.e., anorexia and bulimia), bipolar disorder; developmental or organic mental disorders; and current (past 6 months) substance use disorders and current post-traumatic stress disorder as assessed by clinician at screening visit
* A serious medical condition that may result in surgery or hospitalization.
* A history of head trauma causing prolonged loss of consciousness, or ongoing cognitive impairment
* Inability to understand study procedures or informed consent process, or significant personality dysfunction likely to interfere with study participation (assessed during the clinical interview).
* Subjects who will be non-compliant with the study procedures. This may include planned travel out of town.
* Subjects taking some psychiatric medication such as barbiturates or antipsychotics. Sleep medications and some anti-depressants will be allowed, if the subject has been taken at stable dose 8 weeks prior to baseline and the patient plans to continue at the same dose through the trial.
* Concurrent psychotherapy initiated within 1 month of screen interview, or ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety (such as Cognitive Behavioral Therapy).
* Individuals who have completed a course of MSC or an equivalent meditation training in the last year.
* Individuals reporting significant active suicidal ideation or suicidal behaviors within the past year.
* Individuals with a medical condition (i.e., epilepsy) that may be exacerbated by study treatment, as determined by a study physician or nurse practitioner based on history, physical, and/or labs.
* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-Critical Rumination Scale (SCRS) | 8 weeks
  10-item questionnaire that measures ruminative processes related to self-critical thoughts.
Hospital Anxiety and Disease Scale (HADS) | 8 weeks
  Self-report questionnaire of anxiety and depression symptoms, 14 items using 4-point likert scale

SECONDARY OUTCOMES:
PROMIS Depression Short Form | 8 weeks
  8-item questionnaire that assesses the pure domain of depression in individuals aged 18 and older.
Difficulties in Emotion Regulation Scale-Short Form | 8 weeks
  18-item self-report measure that has established validity and is widely used for assessing emotion regulation style in adults
Penn State Worry Questionnaire (PSWQ) | 8 weeks
  A patient-report measure that is used to understand patients' anxiety, and worry.
PROMIS Anxiety Short Form | 8 weeks
  8 items to assess self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness).
PROMIS Sleep-Anxiety measure | 8 weeks
  13 items from the PROMIS Sleep Disturbance battery, that relate specifically to sleep disturbance resulting from worry, anxiety, or stress.
Liebowitz Social Anxiety Scale (LSAS) | 8 weeks
  A questionnaire widely used to measure social anxiety through situation-based questions that also distinguishes between fear and avoidance ratings.
Self-Compassion Scale (SCS) | 8 weeks
  26-item self-report instrument that uses a 5-point Likert scale for each item to assess compassion and kindness towards oneself, partially through seeing one's experiences as not unique and specific to the individual, but part of a larger human experience.
Fear of Compassion | 8 weeks
  A questionnaire that is the sum of three subscales designed to assess individuals: Compassion for the self-comprised; compassion from others comprised; and compassion for others comprised. We will use the Compassion for Self subscale.
Guilt and Shame Questionnaire (GSQ) | 8 weeks
  8-item survey and is currently the most reliable, valid, and quick-to-complete shame scale for use in therapy outcome studies.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hoge, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Individual-level participant data collected will not be made available to the general public due to conditions of ethical approval regarding confidentiality.